CLINICAL TRIAL: NCT06018766
Title: A Randomized, Placebo-controlled Phase 2 Study to Demonstrate the Safety and Efficacy of the Addition of LAM-001 to Standard Immunosuppression Therapy for Chronic Lung Allograft Dysfunction (BOS).
Brief Title: LAM-001 in Lung Transplant Recipients With Bronchiolitis Obliterans Syndrome.
Acronym: INSPO-BOS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Steven Hays, MD (Other)
Collaborators: OrphAI Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Steven Hays, MD, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAM-001-BOS-CLN01
Record Dates: First submitted 2023-06-01; First posted 2023-08-31 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Bronchiolitis Obliterans Syndrome; Chronic Lung Allograft Dysfunction; Lung Transplantation
Keywords: Bronchiolitis Obliterans Syndrome; Chronic Lung Allograft Dysfunction; Lung Transplant Rejection; Sirolimus; mTOR inhibitor; CLAD
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LAM-001 (Experimental)
  Interventions: Drug: LAM-001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LAM-001 — LAM-001 administered via dry powder inhaler
  Arms: LAM-001
Drug: Placebo — Placebo administered via dry powder inhaler
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn about the safety and effectiveness of LAM-001 in patients who have developed bronchiolitis obliterans syndrome (BOS), a form of chronic rejection, after lung transplantation.

The main questions it aims to answer are:

* Is LAM-001 safe in these patients?
* Is LAM-001 effective in slowing BOS progression?

Participants will:

* Be randomly assigned to inhale either LAM-001 or placebo (a look-alike substance that contains no active drug) daily for 48 weeks
* Attend 10 study visits (mixture of in-person and telehealth) over the 48 week period
* Undergo pulmonary function testing, bronchoscopy, lab testing, and physical examination
* Submit weekly home spirometry monitoring

Researchers will compare participants assigned to LAM-001 versus placebo to see if LAM-001 is safely tolerated and to assess the effectiveness of LAM-001 on slowing BOS progression.

DETAILED DESCRIPTION:
Chronic rejection, commonly denoted as bronchiolitis obliterans (BO), obliterative bronchiolitis (OB), or bronchiolitis obliterans syndrome (BOS), is the leading cause of death beyond the first year after lung transplantation. Whereas the development of BOS is rare within the first year after lung transplantation, annual increments of approximately 10% are recorded in subsequent years, resulting in a cumulative incidence range of 40-50% within the first five years and 70-80% within 10 years of transplantation.

No current effective treatment for BOS exists. BOS represents the leading cause of morbidity and mortality after lung transplantation, limiting 5-year survival to well below other solid organ transplants. BOS is characterized by an inexorable lung function decline despite currently available immunomodulatory treatments. Sirolimus has been shown to block T-cell proliferative effects induced by cytokines, alloantigens, and mitogens in a dose-dependent manner(4, 5). Oral sirolimus has been shown in small studies to have a beneficial impact on rapidly progressive BOS; however, administration in this patient population has been challenged by a high degree of intolerance with the side effects. The development of LAM-001 for lung transplant related BOS, conceptually a T-cell driven process against transplanted alloantigen, is based on the principal hypothesis that administration of a sirolimus dose to the rejecting lung allograft(s) by inhalation will result in improved efficacy by depositing higher drug concentrations directly within the allograft by inhalation than would be achieved by oral administration due to systemic toxicities associated with oral sirolimus. Because of known reduced systemic bioavailability of LAM-001 compared to oral sirolimus dosing, amelioration of the substantial adverse event profile compared to oral drug is expected. LAM-001 is also expected to reduce serious complication risks by obviating requirements for maintenance and augmented immune drugs used to treat BOS.

The primary objective is to assess the clinical efficacy of LAM-001 in lung transplant recipients with bronchiolitis obliterans syndrome as measured by progression free survival and change in forced expiratory volume in one second (FEV1) over a 48-week period. Another primary objective is to assess the safety and tolerability of LAM-001 in lung transplant recipients with bronchiolitis obliterans syndrome.

Secondary objectives are:

* To determine the impact of LAM-001 on genetic markers of bronchiolitis obliterans syndrome and activation of the mammalian target of rapamycin (mTOR) pathway by measuring chronic lung allograft dysfunction signature gene profiling and mTOR pathway activation in bronchoalveolar lavage fluid
* To determine whether donor-derived cell-free DNA (%ddcfDNA) will predict ongoing injury (versus cessation of BOS progression) by measuring %ddcfDNA in randomized subjects. % ddcfDNA will be correlated with clinical outcome measures of FEV1 change, death, and re-transplantation for both randomized groups.
* To determine the levels of sirolimus in the blood and bronchoalveolar lavage (BAL) fluid, the BAL as a surrogate for levels in the lung.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Recipient of a double pulmonary allograft at least 12 months before study entry
* Subjects with clinically diagnosed CLAD-BOS phenotype (all 3 required)

  * BOS defined as screening FEV1 between 85-51% of the baseline as defined by the 2 highest FEV1 measures at least 3 weeks apart.
  * Diagnosis within 12 months of screening visit.
  * FEV1 decline is persistent as defined by decline sustained for > 30 days.
* Currently receiving Standard Immunosuppression. This is defined as a combination of 3 medications including Prednisone, Mycophenolate or Azathioprine, and Tacrolimus or Cyclosporine. The dosing should be stable for 4 weeks prior to screening.
* Absence of oral sirolimus or everolimus treatment for at least 4 weeks prior to screening based on the half-life and resolution of the tissue effects
* Stable enough to enable routine post-transplant bronchoscopy with BAL and biopsy when indicated
* Capable of understanding the purposes and risks of the study
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to study entry
* Women of childbearing potential if sexually active must agree to using highly effective contraception during study and for 90 days after discontinuation of study treatment
* Women of childbearing potential must refrain from breast feeding or donating eggs for the duration of the study and for 90 days after the last dose of study treatment
* Male participants must agree to use a condom during sexual contact with a female of childbearing potential while participating in the study and for 90 days following discontinuation of investigational product use
* Male participants must refrain from donating sperm for the duration of the study and for 90 days after the last dose of study treatment

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Patients with re-transplantation or currently listed for re-transplantation
* Patients with confirmed other causes for loss of lung function, such as acute infection, acute rejection, restrictive allograft syndrome (CLAD - RAS phenotype, see Protocol Specific Definition), etc.
* Patients with acute antibody-mediated rejection at Screening. In this context, clinically stable patients (as judged by the Investigator) with detectable donor-specific antibodies (DSA) levels at the Screening Visit are eligible for the study
* Active acute bacterial, viral, or fungal infection that has not successfully resolved in at least 4 weeks prior to the Screening Visit. Patients with chronic infection or colonization who are clinically stable as per judgement of the investigator are eligible.
* Mechanical ventilation within 12 weeks prior to the randomization
* Patient has baseline resting oxygen saturation of < 89% on room air or use of supplemental oxygen at rest at screening
* Evidence of functional airway stenosis (i.e., bronchomalacia/ tracheomalacia, airway stents, or airways requiring balloon dilatations to maintain patency) with onset after the initial diagnosis of BOS and ongoing at Screening and/or Baseline Visit
* Known hypersensitivity to sirolimus or everolimus
* Currently enrolled in another investigational trial for obstructive chronic lung allograft dysfunction (BOS)
* Patients with chronic renal failure, defined as serum creatinine > 2.5 mg/dL at screening, or requiring chronic dialysis
* Patients with liver disease and serum bilirubin > 3-fold upper limit of normal range or transaminases > 2.5 upper limit of normal range
* Patients with active malignancy within the previous 2 years, including post-transplant lymphoproliferative disorder, except for treated, localized basal and squamous cell carcinomas
* Any history of malignancy likely to result in significant disability or likely to require significant medical or surgical intervention within the next 6 months. This does not include minor surgical procedures for localized skin cancer.
* History of severe allergic reaction to lactose (patients with lactose intolerance are eligible)
* Patients with uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Time to Progression Free Survival (PFS), Level 1 | 52 weeks
  Time to Progression Free Survival (PFS) Level 1, defined as the earliest of the following:
  1. Absolute decrease in FEV1 from baseline of > 10%
  2. Death from respiratory failure

SECONDARY OUTCOMES:
Change in FEV1 | 48 weeks
  Change in FEV1 from baseline
Change in forced expiratory volume in one second/forced vital capacity (FEV1/FVC) | 48 weeks
  Change in FEV1/FVC from baseline
Time to Progression Free Survival (PFS), Level 2 | 52 weeks
  Time to Progression Free Survival (PFS) Level 2, defined as the earliest of the following:
  1. Absolute decrease in the FEV1 from baseline of >20%
  2. Death from respiratory failure

OTHER OUTCOMES:
Change in Quality of Life | 48 weeks
  Change in Quality of Life as measured by St. George's Respiratory Questionnaire -COPD (SGRQ-C). The range of scores is 0-100, with the higher scores representing more limitation in quality of life.
Change in six-minute walk distance (6MWD) | 48 weeks
  Change in 6MWD from baseline
Donor-derived cell-free DNA: Ongoing lung injury | 52 weeks
  Determine whether donor-derived cell-free DNA (%ddcfDNA) will predict ongoing injury (versus cessation of BOS progression) by measuring %ddcfDNA in randomized subjects. %ddcfDNA will be correlated with clinical outcome measures of FEV1 change, death, and re-transplantation for both randomized groups.
% Reduced donor-derived cell-free DNA | 48 weeks
  Determine whether the LAM-001 group will have a salutary effect on allograft injury in terms of reduced %ddcfDNA compared to standard therapy by measuring %ddcfDNA values at determined time points and comparing values between the LAM-001 and placebo groups.
CLAD signature gene profiling | 3 months post randomization
  Utilizing the endobronchial brush, we will quantify a metagene, or normalized sum of gene expression, from our previously published airway inflammation gene set, as described in our publication (PMID: 32885581). The metagene expression will be compared between randomized groups.
mTOR pathway activation | 3 months post randomization
  Utilizing the bronchioalveolar lavage fluid, we will quantify pS6S235/235 in lymphocytes using flow cytometry, to quantify mTORC1 activity, as previously published (PMID: 36066491). We will compare pS6S235/235 between randomized groups.
Blood sirolimus levels | Assessed pre-inhalation at in-person study visits over 48 weeks and post-inhalation at 3 months post randomization
  Measured blood sirolimus levels
Bronchioalveolar lavage fluid sirolimus levels | 12 weeks
  Measured bronchioalveolar lavage fluid sirolimus levels
Airway Hypersensitivity to Treatment | Baseline Study Visit (Week 0)
  Measurement of FEV1 pre-inhalation and 4 hours following study drug inhalation to determine whether a subject has airway hyperreactivity to the study drug.
Adverse events | 52 weeks
  Incidence and severity of treatment emergent adverse events (AE) and serious adverse events (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hays, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillen JR, Zhao Y, Harris DA, LaPar DJ, Kron IL, Lau CL. Short-course rapamycin treatment preserves airway epithelium and protects against bronchiolitis obliterans. Ann Thorac Surg. 2013 Aug;96(2):464-72. doi: 10.1016/j.athoracsur.2013.04.068. Epub 2013 Jun 24. PMID 23806229
- [Background] Gillen JR, Zhao Y, Harris DA, Lapar DJ, Stone ML, Fernandez LG, Kron IL, Lau CL. Rapamycin blocks fibrocyte migration and attenuates bronchiolitis obliterans in a murine model. Ann Thorac Surg. 2013 May;95(5):1768-75. doi: 10.1016/j.athoracsur.2013.02.021. Epub 2013 Apr 2. PMID 23561805
- [Background] Zhao Y, Gillen JR, Meher AK, Burns JA, Kron IL, Lau CL. Rapamycin prevents bronchiolitis obliterans through increasing infiltration of regulatory B cells in a murine tracheal transplantation model. J Thorac Cardiovasc Surg. 2016 Feb;151(2):487-96.e3. doi: 10.1016/j.jtcvs.2015.08.116. Epub 2015 Sep 7. PMID 26481278
- [Background] Sehgal SN. Rapamune (RAPA, rapamycin, sirolimus): mechanism of action immunosuppressive effect results from blockade of signal transduction and inhibition of cell cycle progression. Clin Biochem. 1998 Jul;31(5):335-40. doi: 10.1016/s0009-9120(98)00045-9. PMID 9721431
- [Background] Bak S, Tischer S, Dragon A, Ravens S, Pape L, Koenecke C, Oelke M, Blasczyk R, Maecker-Kolhoff B, Eiz-Vesper B. Selective Effects of mTOR Inhibitor Sirolimus on Naive and CMV-Specific T Cells Extending Its Applicable Range Beyond Immunosuppression. Front Immunol. 2018 Dec 17;9:2953. doi: 10.3389/fimmu.2018.02953. eCollection 2018. PMID 30619313
- [Background] Sonis S, Treister N, Chawla S, Demetri G, Haluska F. Preliminary characterization of oral lesions associated with inhibitors of mammalian target of rapamycin in cancer patients. Cancer. 2010 Jan 1;116(1):210-5. doi: 10.1002/cncr.24696. PMID 19862817
- [Background] Boers-Doets CB, Raber-Durlacher JE, Treister NS, Epstein JB, Arends AB, Wiersma DR, Lalla RV, Logan RM, van Erp NP, Gelderblom H. Mammalian target of rapamycin inhibitor-associated stomatitis. Future Oncol. 2013 Dec;9(12):1883-92. doi: 10.2217/fon.13.141. PMID 24295418
- [Background] Vigarios E, Epstein JB, Sibaud V. Oral mucosal changes induced by anticancer targeted therapies and immune checkpoint inhibitors. Support Care Cancer. 2017 May;25(5):1713-1739. doi: 10.1007/s00520-017-3629-4. Epub 2017 Feb 22. PMID 28224235
- [Background] Pilotte AP, Hohos MB, Polson KM, Huftalen TM, Treister N. Managing stomatitis in patients treated with Mammalian target of rapamycin inhibitors. Clin J Oncol Nurs. 2011 Oct;15(5):E83-9. doi: 10.1188/11.CJON.E83-E89. PMID 21951751
- [Background] de Oliveira MA, Martins E Martins F, Wang Q, Sonis S, Demetri G, George S, Butrynski J, Treister NS. Clinical presentation and management of mTOR inhibitor-associated stomatitis. Oral Oncol. 2011 Oct;47(10):998-1003. doi: 10.1016/j.oraloncology.2011.08.009. Epub 2011 Sep 3. PMID 21890398